CLINICAL TRIAL: NCT05072288
Title: A Remote Physical Activity Program Via the PACE Tool to Counter the Physical Impairments, Accentuated by the Pandemic, in the Population Suffering from Type 1 Myotonic Dystrophy
Brief Title: A Remote Physical Activity Program in the Population Suffering from Type 1 Myotonic Dystrophy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-791
Record Dates: First submitted 2021-08-10; First posted 2021-10-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
Keywords: Myotonic dystrophy type 1; Physical activity; function; balance; mobility
MeSH Terms: conditions — Myotonic Dystrophy; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will receive an adapted remote physical program. Half of the participants will do a 12 weeks control prior to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote activity program (Experimental): Activity program based on objective evaluation. Possibility of 35 different programs primarily targeting impairments (lower limb, upper limb or balanced)
  Interventions: Other: Remote activity program

INTERVENTIONS:
Other: Remote activity program — Participant will have to do exercise at home everyday (15min/day)

SUMMARY:
The COVID-19 pandemic exacerbates health problems by reducing access to adapted and advanced physical rehabilitation for several people who need rehabilitation services, including the population with myotonic dystrophy type 1 (DM1). The PACE tool, an innovative web tool integrating pragmatic physical activity programs, seems to be an interesting and innovative intervention to counter physical deficiencies of people with DM1, which are unfortunately accentuated by the pandemic, while reducing the risk of COVID-19 exposure. Objectives: 1) Evaluate the feasibility, usability and acceptability of the PACE tool in the DM1 population; 2) Evaluate the effects of the intervention on their physical and cognitive health; and 3) Estimate the cost-effectiveness ratio of this intervention. Method: Sixty people (experimental group = 40 and control group = 20) will participate in this randomized intervention study. Participants in the experimental group will be assigned to one of the 35 physical activity programs adapted to their condition of the PACE tool. The program must be performed on a daily basis for a period of 12 weeks. Physical and cognitive health will be assessed before and after the remote intervention via ZOOM, for all participants.

ELIGIBILITY:
Inclusion Criteria:

* DM1 diagnosis must be confirmed by genetic analysis (juvenile, adults or late-onset phenotypes);
* Aged between 18 and 60 years old;
* Be able to do exercise;
* Subjects must be able to give their consent freely and voluntarily.

Exclusion Criteria:

* Patients who already train (>3 times per week or >150min/week);
* Don't speak french or english;
* Are not able to do exercise (even in sitting position);

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Functional capacity from baseline to week 12 | Week 12
  Short physical performance battery Functional reach test
Change in the Level of physical activity from baseline to week 12 | Week 12
  Rapid Assessment of physical Activity & International Physical Activity Questionnaires
Feasability/acceptability of the program and Satisfaction | Week 12
  Number of sessions completed/planned Likert System Usability Scale.

SECONDARY OUTCOMES:
Changes in the score of the Fatigue and Daytime Sleepiness Scale from baseline to week 12 | Week 12
  Changes in the score of the Fatigue and Daytime Sleepiness Scale (FDSS). The FDSS is a 12-item questionnaire where all questions are scored from 0 to 2. A higher score means more daytime sleepiness and fatigue.
Changes in the Marin apathy scale from baseline to week 12 | Week 12
  Changes in the Marin apathy scale. The Marin apathy scale is scored by the clinician where he interviews the subject and then scores an 18-item list on a scale of 1 to 4. A high score means more apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Duchesne, Principal Investigator — Université du Québec à Chicoutimi
Locations (2):
- Canada (2):
  - Groupe de recherche interdisciplinaire Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Jonquière, Quebec
  - Université du Québec à Chicoutimi, Saguenay, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouchard G, Roy R, Declos M, Mathieu J, Kouladjian K. Origin and diffusion of the myotonic dystrophy gene in the Saguenay region (Quebec). Can J Neurol Sci. 1989 Feb;16(1):119-22. doi: 10.1017/s0317167100028651. PMID 2924205
- [Background] Mateos-Aierdi AJ, Goicoechea M, Aiastui A, Fernandez-Torron R, Garcia-Puga M, Matheu A, Lopez de Munain A. Muscle wasting in myotonic dystrophies: a model of premature aging. Front Aging Neurosci. 2015 Jul 9;7:125. doi: 10.3389/fnagi.2015.00125. eCollection 2015. PMID 26217220
- [Background] Gagnon C, Petitclerc E, Kierkegaard M, Mathieu J, Duchesne E, Hebert LJ. A 9-year follow-up study of quantitative muscle strength changes in myotonic dystrophy type 1. J Neurol. 2018 Jul;265(7):1698-1705. doi: 10.1007/s00415-018-8898-4. Epub 2018 May 21. PMID 29785524
- [Background] Petitclerc E, Hebert LJ, Mathieu J, Desrosiers J, Gagnon C. Lower limb muscle strength impairment in late-onset and adult myotonic dystrophy type 1 phenotypes. Muscle Nerve. 2017 Jul;56(1):57-63. doi: 10.1002/mus.25451. Epub 2016 Nov 25. PMID 27784130
- [Background] Petitclerc E, Hebert LJ, Mathieu J, Desrosiers J, Gagnon C. Relationships between Lower Limb Muscle Strength Impairments and Physical Limitations in DM1. J Neuromuscul Dis. 2018;5(2):215-224. doi: 10.3233/JND-170291. PMID 29865087
- [Background] Hammaren E, Kjellby-Wendt G, Lindberg C. Muscle force, balance and falls in muscular impaired individuals with myotonic dystrophy type 1: a five-year prospective cohort study. Neuromuscul Disord. 2015 Feb;25(2):141-8. doi: 10.1016/j.nmd.2014.11.004. Epub 2014 Nov 13. PMID 25475393
- [Background] Wiles CM, Busse ME, Sampson CM, Rogers MT, Fenton-May J, van Deursen R. Falls and stumbles in myotonic dystrophy. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):393-6. doi: 10.1136/jnnp.2005.066258. Epub 2005 Sep 30. PMID 16199443
- [Background] Gallais B, Montreuil M, Gargiulo M, Eymard B, Gagnon C, Laberge L. Prevalence and correlates of apathy in myotonic dystrophy type 1. BMC Neurol. 2015 Aug 22;15:148. doi: 10.1186/s12883-015-0401-6. PMID 26296336
- [Background] Gagnon C, Mathieu J, Jean S, Laberge L, Perron M, Veillette S, Richer L, Noreau L. Predictors of disrupted social participation in myotonic dystrophy type 1. Arch Phys Med Rehabil. 2008 Jul;89(7):1246-55. doi: 10.1016/j.apmr.2007.10.049. PMID 18586127
- [Background] Bertran Recasens B, Rubio MA. Neuromuscular Diseases Care in the Era of COVID-19. Front Neurol. 2020 Nov 26;11:588929. doi: 10.3389/fneur.2020.588929. eCollection 2020. PMID 33329336
- [Background] Di Stefano V, Battaglia G, Giustino V, Gagliardo A, D'Aleo M, Giannini O, Palma A, Brighina F. Significant reduction of physical activity in patients with neuromuscular disease during COVID-19 pandemic: the long-term consequences of quarantine. J Neurol. 2021 Jan;268(1):20-26. doi: 10.1007/s00415-020-10064-6. Epub 2020 Jul 13. PMID 32661716
- [Background] Carvalho LP, Kergoat MJ, Bolduc A, Aubertin-Leheudre M. A Systematic Approach for Prescribing Posthospitalization Home-Based Physical Activity for Mobility in Older Adults: The PATH Study. J Am Med Dir Assoc. 2019 Oct;20(10):1287-1293. doi: 10.1016/j.jamda.2019.01.143. Epub 2019 Mar 11. PMID 30872083
- [Background] Fruteau de Laclos L, Sirois MJ, Blanchette A, Martel D, Blais J, Emond M, Daoust R, Aubertin-Leheudre M. Exercise Interventions for Community-Dwelling Older Adults Following an Emergency Department Consultation for a Minor Injury. J Aging Phys Act. 2021 Apr 1;29(2):267-279. doi: 10.1123/japa.2019-0200. Epub 2020 Oct 27. PMID 33108761
- [Background] Aubertin-Leheudre M, Rolland Y. The Importance of Physical Activity to Care for Frail Older Adults During the COVID-19 Pandemic. J Am Med Dir Assoc. 2020 Jul;21(7):973-976. doi: 10.1016/j.jamda.2020.04.022. Epub 2020 Apr 30. No abstract available. PMID 32513558
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Hilgers RD, Roes K, Stallard N; IDeAl, Asterix and InSPiRe project groups. Directions for new developments on statistical design and analysis of small population group trials. Orphanet J Rare Dis. 2016 Jun 14;11(1):78. doi: 10.1186/s13023-016-0464-5. PMID 27301273